CLINICAL TRIAL: NCT04078958
Title: Health Effects of Salmon Fish Meal - ex Vivo Study
Brief Title: Effects of Salmon Fishmeal Ex Vivo (FishMeal Ex Vivo)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Kirsten Holven, Professor, University of Oslo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019/875/REK sør-øst B
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Metabolic Disease; Inflammation; Endocrine; Obesity
MeSH Terms: conditions — Metabolic Diseases; Inflammation; Obesity | interventions — Whey

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salmon fishmeal (Experimental): 5 g fishmeal in capsules, single oral dose
  Interventions: Dietary Supplement: Salmon fishmeal
- Whey (Active Comparator): 5 g whey in capsules, single oral dose
  Interventions: Dietary Supplement: Whey

INTERVENTIONS:
Dietary Supplement: Salmon fishmeal — Salmon fishmeal with high protein content
  Arms: Salmon fishmeal
Dietary Supplement: Whey — Whey with high protein content
  Arms: Whey

SUMMARY:
Diabetes contributes significantly to the burden of disease in Norway and cardiovascular disease is the main cause of mortality.

Both lean and fatty fish are shown to have beneficial health effects. In addition to omega-3 fatty acids, fish contain potential health-promoting components such as taurine, vitamin D, vitamin B12, iodine, selenium and more unspecified components such as bioactive peptides. With the expected growth in the aquaculture sector, more protein-rich by-products will become available.

The overall aim of this project is to investigate physiological and molecular effects of fish protein in the form of salmon fishmeal compared to whey in a human intervention study with regard to carbohydrate- and fat metabolism, endocrine factors and inflammation.

The investigators will include healthy subjects to a randomized controlled cross over study. The subjects will receive a single, oral dose of fishmeal or whey. Blood samples are taken before (fasting) and 30 and 60 minutes after intake. The molecular effects of fishmeal and whey are investigated ex vivo. This is done by incubating human cell lines (i.e hepatocytes, adipocytes, epithelial cells) with fasting and postprandial serum from the participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.5-24.9 kg/m2

Exclusion Criteria:

* Body mass index <18.5 or >24.9 kg/m2
* Known diabetes or high blood pressure
* Pregnancy or breast feeding
* Allergy or intolerance to dairy or fish/fish protein.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Changes in the whole genome transciptome in cultured cells | Acute changes from baseline to 30 and/or 60 minutes.
  Changes in the whole genome transciptome of cultured cells incubated with fasting and postprandial serum from participants receiving whey or fishmeal.

SECONDARY OUTCOMES:
Changes in histone marks on selected target genes in cultured cell lines | Acute changes from baseline to 30 and/or 60 minutes.
  Changes in histone marks on selected target genes in cultured cells incubated with fasting or postprandial serum from participants receiving whey or fishmeal.
Changes in insulin-stimulated glucose uptake in cultured cell lines | Acute changes from baseline to 30 and/or 60 minutes.
  Changes in insulin sensitivity measured as insulin-stimulated glucose uptake of cultured cells incubated with fasting and postprandial serum from participants receiving whey or fishmeal.
Changes in cytokine secretion in cultured cell lines | Acute changes from baseline to 30 and/or 60 minutes.
  Changes in inflammatory and endocrine factors measured as the secretion of single cytokines from cultured cells incubated with fasting and postprandial serum from participants receiving whey or fishmeal. The choice of factors will be guided by the results from the primary endpoint.
Blood concentration of insulin | Acute changes from baseline to 30 and 60 minutes
  Blood concentration of insulin in participants receiving whey or fishmeal.
Blood concentration of glucose | Acute changes from baseline to 30 and 60 minutes
  Blood concentration of glucose in participants receiving whey or fishmeal.
Blood concentration of triglycerides | Acute changes from baseline to 30 and 60 minutes
  Blood concentration of triglycerides in participants receiving whey or fishmeal.
Blood concentration of cholesterol | Acute changes from baseline to 30 and 60 minutes
  Blood concentration of total cholesterol in participants receiving whey or fishmeal.
Markers in blood related to appetite | Acute changes from baseline to 30 and 60 minutes
  Blood concentration of the appetite hormones, i.e. GLP-1, Leptin and GIP in participants receiving whey or fishmeal.
Markers in blood related to low grade inflammation | Acute changes from baseline to 30 and 60 minutes
  Blood concentration of microCRP in participants receiving whey or fishmeal.
Markers in blood related to digestion of protein | Acute changes from baseline to 30 and/or 60 minutes
  Blood concentration of amino acids and small peptides in participants receiving whey or fishmeal.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Holven, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No